CLINICAL TRIAL: NCT01645293
Title: Multicentre Phase I Trial of Engineered T Cells for Patients With Relapsed or Refractory Primary Cutaneous CD30+ Large T Cell Lymphoma or Transformed CD30+ Mycosis Fungoides
Acronym: TECLA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Dr. rer. nat Cornelia Mauch, Consultant dermatologist, CIO tumor centre, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1065
Record Dates: First submitted 2012-07-11; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: CD30 Positive Cutaneous T Cell Lymphoma; CD30 Positive Transformed Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genetically modified T cells #1138 (Experimental)
  Interventions: Genetic: Genetically modified T cells # 1138

INTERVENTIONS:
Genetic: Genetically modified T cells # 1138

SUMMARY:
Patients with cutaneous CD30 positive lymphoma will receive systemical and topical treatment with their own genetically modified T cells. Treatment evaluation consists of assessment of safety and preliminary evidence of response.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent, prior to pre-study screening and treatment, with the understanding that the consent may be withdrawn by the patient at any time without prejudice, ability to understand the written informed consent document.
* Male or female > 18 years of age to 70 years of age
* Diagnosis of primary cutaneous CD30+ large T cell lymphoma OR
* Diagnosis of transformed CD30+ mycosis fungoides, i.e.,
* Histological confirmation of diagnosis.
* multiple (> 5) cutaneous tumor lesions (TNM EORTC 2007 T3, N1, clinical stage <IIb),
* Measurable disease according to RECIST criteria
* Refractory or relapsed disease after at least one line of treatment, e.g. PUVA (Psoralen plus UVA), PUVA + Interferon, oral Bexarotene, low dose MTX)
* ECOG performance status 0-3
* Life expectancy > 12 months
* Female patients with childbearing potential must have a negative serum pregnancy test within two weeks of first dose of study drug. Male and female patients must agree to use an effective oral contraceptive method while on study treatment, if appropriate, and for a minimum of twelve months following study therapy

Exclusion Criteria:

* Previously untreated patients
* Presence of any organ or brain involvement as determined during tumor staging by contrast computed tomography [CT] or magnetic resonance imaging [MRI] scan
* Known hereditary blood coagulation disorders/DIC
* Prior allogeneic hematopoietic stem-cell or organ transplantation
* Severe cardiovascular disease like functionally restricting heart rhythm disturbance or heart malformation or severe hypertension, or cardiac insufficiency > NHYA-II
* known active infection including HIV, Hepatitis B or C, VZV, or CMV
* Insufficient bone marrow reserve (Leucocytes <3.500/μl; Thrombocytes <100.000/μl)
* Creatinine-Clearance < 50 ml/min or Crea > 1.8 mg/dl
* Bilirubin > 2 mg/dl; ASAT, ALAT > 2.5xN
* Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
* Known pulmonary dysfunction
* Requirement of chronic immune suppression
* Treatment with corticosteroids for concomitant or intercurrent disease
* Having participated in another clinical trial or any IND in the preceding 4 weeks
* Anti-cancer chemotherapy in the preceding 4 weeks
* Known drug abuse/alcohol abuse
* Known allergic/hypersensitivity reaction to any of the components of the treatment
* Known serious uncontrolled infections
* Known active secondary malignancy or other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the skin or cervix
* Medical or psychological condition or inadequate knowledge of german language which in the opinion of the investigator would not permit the patient to complete the study or meaningfully sign informed consent
* Legal incapacity or limited legal capacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)

PRIMARY OUTCOMES:
Rate of patients experiencing dose limiting toxicities of engineered T cells #1138.
Definition of maximum tolerated dose (MTD) of engineered T cells #1138.

SECONDARY OUTCOMES:
Preliminary evidence of response to treatment
  * Complete Response (CR): Disappearance of treated lesion.
  * Partial Response (PR): At least 30% decrease in the sum of two diameters compared to the initiatal diameters of the treated lesion.
  * Progressive Disease (PD): At least 20% increase in the sum of two diameters of treated lesions.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of two diameters while on study.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, Germany